CLINICAL TRIAL: NCT00006127
Title: Phase I Study of Amifostine in Patients With Bone Marrow Failure Related to Fanconi's Anemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dana-Farber Cancer Institute (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/15281; DFCI-9910170; ALZA-99-004-ii
Record Dates: First submitted 2000-08-03; First posted 2000-08-04 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-10

CONDITIONS: Fanconi's Anemia
Keywords: Fanconi's anemia; aplastic anemia; hematologic disorders; rare disease
MeSH Terms: conditions — Fanconi Anemia; Anemia, Aplastic; Hematologic Diseases; Rare Diseases | interventions — Amifostine

INTERVENTIONS:
Drug: amifostine

SUMMARY:
OBJECTIVES:

I. Evaluate the toxicity of amifostine in patients with bone marrow failure related to Fanconi's anemia.

II. Determine the efficacy of this treatment regimen in this patient population.

III. Evaluate the effect of this treatment regimen on bone marrow progenitor cell proliferation and peripheral blood mononuclear cell apoptosis in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a dose escalation study.

Patients receive amifostine IV over 3-5 minutes three times a week for three weeks.

Cohorts of 3 patients receive one of three dose levels of amifostine. The maximum tolerated dose is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed weekly for 3 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of Fanconi's anemia by conventional diepoxybutane or mitomycin sensitivity assays, or molecular testing

Bone marrow failure verified on at least 3 occasions in the preceding 3 months by any one of the following: hemoglobin less than 8 g/dL; absolute neutrophil count less than 1,000/mm3; platelet count less than 30,000/mm3; symptomatic bone marrow failure (e.g., exercise limitation from anemia or spontaneous bleeding from thrombocytopenia)

Evidence consistent with myelodysplastic syndrome allowed if less than 5% blasts on bone marrow aspiration; clonality on bone marrow cytogenetic analysis OR morphological changes on bone marrow aspirate

Refusal of or unsuccessful with prior conventional therapies

--Prior/Concurrent Therapy--

Biologic therapy: No prior bone marrow transplantation; no concurrent hematopoietic growth factors

Endocrine therapy: No concurrent androgens

--Patient Characteristics--

Hepatic: Bilirubin no greater than 2 times normal AST no greater than 3 times normal ALT no greater than 6 times normal

Renal: Creatinine no greater than 2 times normal

Other: No prior malignancy; no active bacterial, viral, or fungal infection requiring therapy other than prophylaxis; not pregnant; negative pregnancy test

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: W. Nicholas Haining, Study Chair — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States